CLINICAL TRIAL: NCT00429975
Title: Comparison Between Ceftriaxone and Levofloxacin on Cytokine Expression Over Time in Severe Pneumococcal Pneumonia
Brief Title: Ceftriaxone Vs Levofloxacin on Cytokine Expression in Pneumococcal Pneumonia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIS G03/103
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Pneumonia, Pneumococcal
Keywords: fluorquinolones,; b-lactams,; immunomodulation.
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — Levofloxacin; Ceftriaxone

INTERVENTIONS:
Drug: levofloxacin
Drug: ceftriaxone

SUMMARY:
The purpose of this study is to compare levofloxacin vs ceftriaxone impact on the cytokine production in patients with pneumococcal pneumonia.

DETAILED DESCRIPTION:
Bacterial alveolar invasion is followed by a compartmentalized inflammatory response. Data suggest that some antimicrobials may induce a differential release of cytokines, with the potential of either accelerating or down regulating cytokine production.

The aim of our study was to compare the effects of ceftriaxone compared with levofloxacin on cytokine systemic concentrations in patients with pneumococcal pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* patients with an acute febrile respiratory illness accompanied by a new radiographic infiltrate consistent with this diagnosis.
* and with a confirmed pneumococcal aetiology

Exclusion Criteria:

* age < 18 years,
* pneumonia distal to endobronchial obstruction,
* pulmonary tuberculosis,
* bronchiectasis,
* known allergy to B-lactams or fluoroquinolones,
* underlying systemic autoimmune disease
* immunocompromised states including patients on maintenance oral corticosteroids, HIV infection,
* pregnancy,
* patients that received antimicrobial therapy in the 15 days preceding the current episode and those who had received fluoroquinolones in the last month, or non steroidal anti-inflammatory therapy in the last two weeks.
* Patients with renal failure (serum creatinine > 2 mg / dL),
* and patients with a documented pneumococcal pneumonia in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-08; Study Completion 2005-09

PRIMARY OUTCOMES:
Circulating levels of pro and anti-inflammatory cytokines at 0h, 24, 72 h and 120 h from inclusion

SECONDARY OUTCOMES:
the relationship between cytokine expression, clinical variables and severity of disease.

CONTACTS AND LOCATIONS:
Overall Officials: ESTHER CALBO, MD, Principal Investigator — Hospital Mutua de Terrassa; MONTSERRAT ALSINA, MD, Principal Investigator — HOSPITAL MUTUA TERRASSA; MARIONA XERCAVINS, MD, Principal Investigator — Hospital Mutua de Terrassa; EVA CUCHI, MD, Principal Investigator — Hospital Mutua de Terrassa; MONICA RODRIGUEZ-CARBALLEIRA, PhD, Principal Investigator — Hospital Mutua de Terrassa; JAVIER GARAU, PhD, Study Director — Hospital Mutua de Terrassa
Locations (1):
- Hospital Mutua de Terrassa, Terrassa, BARCELONA, Spain